CLINICAL TRIAL: NCT04523779
Title: A Pragmatic Trial of Brief CBT for Anxiety in VA Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 18-233; HX-002796 (Other Grant/Funding Number: VA Health Services Research); CIRB 20-22 (Other: VA Central Institutional Review Board)
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
Keywords: anxiety disorder; panic disorder; phobia, social; worry; stress
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Phobia, Social

STUDY DESIGN:
Intervention Model Description: Cognitive behavioral therapy (CBT) is an evidence-based practice (EBP) for all types of anxiety disorders including generalized anxiety disorder (GAD), panic disorder, and social anxiety disorder. The proposed bCBT treatment for anxiety was specifically designed for use within VA PCMHI settings and uses a patient-centered approach to increase engagement while addressing the mental health needs of anxious Veterans. Emphasis was placed on maximizing intervention potency and minimizing intensity and duration to improve implementation value and alignment with VA PCMHI requirements. The intervention directly addresses challenges to delivery of CBT providing 1) a brief, practical model of care to address multiple anxiety conditions consistent with the PCMHI model (e.g. 4-6 sessions; measurement-based care), and 2) a clinically potent intervention that includes exposure-based skills.
Who Masked: Outcomes Assessor
Masking Description: Outcome data will be collected by independent evaluators (IEs) who will be blinded to randomization. All IEs will be based in Houston, with direct oversight by Dr. Cully. IEs will undergo training and calibration on all study measures and be regularly reassessed for quality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Cognitive Behavioral Therapy (Experimental): The proposed bCBT treatment for anxiety was specifically designed for use within VA PCMHI settings and uses a patient-centered approach to increase engagement while addressing the mental health needs of anxious Veterans. Emphasis was placed on maximizing intervention potency and minimizing intensity and duration to improve implementation value and alignment with VA PCMHI requirements. The intervention directly addresses challenges to delivery of CBT providing 1) a brief, practical model of care to address multiple anxiety conditions consistent with the PCMHI model (e.g. 4-6 sessions; measurement-based care), and 2) a clinically potent intervention that includes exposure-based skills.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy
- Enhanced Usual Care (No Intervention): EUC participants will receive anxiety education materials, a note in their medical record indicating the presence of elevated anxiety symptoms, and 4 brief monthly check-in calls with project staff. The primary outcome, anxiety symptoms, will be evaluated at 4-, 8- and 12-month follow-ups. Due to ethical concerns of withholding needed treatment, EUC participants will NOT be restricted from receiving mental health services including psychotherapy during the study period. The investigators fully expect that EUC participants may receive anxiety treatments (e.g., antianxiety and antidepressant medications or psychotherapy).

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy — The proposed bCBT treatment for anxiety was specifically designed for use within VA PCMHI settings and uses a patient-centered approach to increase engagement while addressing the mental health needs of anxious Veterans. Emphasis was placed on maximizing intervention potency and minimizing intensity and duration to improve implementation value and alignment with VA PCMHI requirements. The intervention directly addresses challenges to delivery of CBT providing 1) a brief, practical model of care to address multiple anxiety conditions consistent with the PCMHI model (e.g. 4-6 sessions; measurement-based care), and 2) a clinically potent intervention that includes exposure-based skills.
  Other Names: bCBT
  Arms: Brief Cognitive Behavioral Therapy

SUMMARY:
This 4-year study will examine the value of a type of a brief cognitive behavioral therapy treatment for Veterans with anxiety and worry. This treatment will be delivered either in-person, or by video telehealth to the Veteran's home. The treatment will be delivered by providers at three Veterans Administration Medical Centers (Houston, New Orleans, and San Antonio). The study will compare the helpfulness of this treatment to the usual care Veterans receive for anxiety and worry. A supplement to this study will also evaluate daily discrimination experiences of Veterans based on the participant's race, ethnicity, religion, physical appearance, or other characteristics.

DETAILED DESCRIPTION:
This 4-year, multisite trial (Houston, New Orleans and San Antonio) will use a pragmatic randomized trial design to examine the effectiveness and implementation potential of a brief cognitive behavioral therapy(bCBT) intervention for anxiety delivered either in-person or via VA Video Connect-Home (VVC-H), according to patient preference. Brief CBT will be delivered by existing Primary Care Mental Health Integration (PCMHI) providers at three large VAMCs (Houston, New Orleans, and San Antonio). Aim 1 will examine the clinical effectiveness of the bCBT intervention vs. Enhanced Usual Care (EUC) for anxiety at 4-, 8-, and 12-month follow-ups. Aim 2 will determine factors associated with bCBT response and explore Veteran demographic and clinical factors associated with VVC-H engagement. An exploratory aim will use mixed, qualitative and quantitative methods to better understand implementation successes and challenges related to delivery and impact of bCBT anxiety and VVC-H use in the PCMHI setting. The primary hypothesis is that anxiety outcomes, as measured by the General Anxiety Disorder 7-item scale (GAD-7) will be superior at 4-, 8-, and 12-month follow up for patients who are assigned to receive bCBT vs. EUC.

In addition, participants will be asked to complete the Diversity Supplement measures and qualitative interview to evaluate whether sociocultural factors are associated with the severity and type of anxiety symptoms among Veterans of different race/ethnicity groups.

ELIGIBILITY:
Inclusion Criteria:

* Must be a United States military Veteran
* Veteran participants will be current recipients of services at the Houston, New Orleans, or San Antonio VA Medical Centers.
* Patients who have received Primary Care Mental Health Integration services, or are eligible for PCMHI services (They are not receiving specialty mental health services)
* Veterans with clinically significant symptoms of anxiety will be included after screening on two occasions to ensure consistency of anxiety symptoms (GAD-7 score of 10 or greater; telephone screen and baseline appointment).

Exclusion Criteria:

* Cognitive impairment
* Presence of bipolar, psychotic or substance-abuse disorders.
* Veterans currently receiving psychotherapy for anxiety at the time of enrollment WILL be excluded so as not to duplicate services (Current treatment will be defined as patients that have received a psychotherapy appointment within the last 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
GAD-7 Change | Baseline, 4-, 8-, and 12-month
  The GAD-7 is a seven-item self-report instrument for screening, diagnosis and severity assessment of anxiety disorder. It is psychometrically strong and valid for use in the primary care setting. A GAD-7 score of 10 or higher will be required for study inclusion. Treatment response will be defined as a 50% reduction in baseline GAD-7 scores. The GAD-7 total score for the seven items ranges from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.

SECONDARY OUTCOMES:
OASIS Change | Baseline, 4-, 8-, and 12-month
  The Overall Anxiety Severity and Impairment Scale (OASIS) will be a secondary measure of anxiety. Unlike the GAD-7, which will be administered by both research staff and PCMHI providers, the OASIS will only be administered by research staff, thereby avoiding response bias that may occur in the clinical setting. The OASIS is a widely used five-item measure of anxiety for primary care settings assessing anxiety frequency, anxiety severity, avoidance behaviors, social interference, and interference at work, school, or home. Each item of the OASIS instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4 and can be summed to obtain a total score ranging from 0 to 20. A higher score indicates a poorer outcome.
SF-12 Change | Baseline, 4-, 8-, and 12-month
  The SF-12 is a self-reported outcome measure assessing the impart of health on an individual's everyday life. Physical and Mental Health Composite Scores are computed using the score of 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The investigators will assess quality of life using the 12-item Short Form Health Survey for Veterans (SF-12V18), an instrument adopted by VHA as a measure of functional status. SF-12V responses can be summarized in component scores for physical (PCS) and mental (MCS) functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Terri L. Fletcher, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (3):
- United States (3):
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cully JA, Fischer EP, Gonzalez R, Williams JS, Sansgiry S, Zeno D, Mittal D, Kuo I. Provider perceptions and use of mental health services in the Veterans Health Administration during the COVID-19 pandemic. Psychol Serv. 2024 Feb;21(1):110-119. doi: 10.1037/ser0000772. Epub 2023 Jun 1. PMID 37261762
- [Background] Ecker AH, Cully JA, Cucciare MA, Hundt NE. Patient and Provider Perspectives on Treating Substance Use Disorder and Co-Occurring Anxiety and Posttraumatic Stress Disorders in the Veterans Affairs Healthcare System. Journal of Veterans Studies. 2023 Jun 1; 9(1):171-180.
- [Background] Cully JA, Hundt NE, Fletcher T, Sansgiry S, Zeno D, Kauth MR, Kunik ME, Sorocco K. Brief Cognitive-Behavioral Therapy for Depression in Community Clinics: A Hybrid Effectiveness-Implementation Trial. Psychiatr Serv. 2024 Mar 1;75(3):237-245. doi: 10.1176/appi.ps.20220582. Epub 2023 Sep 7. PMID 37674395
- [Background] Hertz AG, Dawson DB, Rassu FS, Ecker AH, Helm A, Hundt NE, Fletcher TL. Delivery of Exposure and Response Prevention Among Veterans with Obsessive-Compulsive Disorder. J Behav Health Serv Res. 2023 Oct;50(4):514-523. doi: 10.1007/s11414-023-09838-3. Epub 2023 Apr 6. PMID 37024645
- [Background] Boykin DM, Wray LO, Funderburk JS, Holliday S, Kunik ME, Kauth MR, Fletcher TL, Mignogna J, Roberson RB 3rd, Cully JA. Leveraging the ExpandNet framework and operational partnerships to scale-up brief Cognitive Behavioral Therapy in VA primary care clinics. J Clin Transl Sci. 2022 Jul 20;6(1):e95. doi: 10.1017/cts.2022.430. eCollection 2022. PMID 36003211

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04523779/ICF_000.pdf